CLINICAL TRIAL: NCT06970834
Title: Using Continuous Glucose Monitoring Tools to Explore the Effect of Bitter Melon Peptides on Glycemic Control and Metabolic Indicators in Diabetic Patients
Brief Title: Explore the Effect of Bitter Melon Peptides on Glycemic Control and Metabolic Indicators in Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, PEI-YUNG LIAO, Chief of Division of Endocrinology and Metabolism, Department of Internal Medicine, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCH IRB 250121
Record Dates: First submitted 2025-04-24; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Diabetes
Keywords: bitter melon peptides
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A total of 160 diabetic patients on Metformin monotherapy will be recruited and randomized into either the bitter melon peptide group or the placebo group for a 12-week clinical intervention
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bitter melon peptides (Experimental): Bitter melon peptide contains various active substances such as bitter melon saponins and bitter melon polysaccharides.
  Interventions: Dietary Supplement: bitter melon peptides
- Placebo group (Placebo Comparator): The placebo capsule containing microcrystalline cellulose. The placebo is identical in appearance, color, and dosage schedule to the intervention product, but does not contain any active ingredients.
  Interventions: Dietary Supplement: bitter melon peptides

INTERVENTIONS:
Dietary Supplement: bitter melon peptides — Momordica charantia extract

SUMMARY:
The goal of this clinical trial is to learn the potential of bitter melon peptides in stabilizing blood glucose in diabetic adults. It will also learn about the effects of bitter melon peptides on metabolic parameters. The main questions it aims to answer are:

* the regulatory effects of bitter melon peptides on glycemic variability
* impact on glycemic and metabolic indicators Researchers will compare bitter melon peptides to a placebo (a look-alike capsule that contains Microcrystalline Cellulose) to see if bitter melon peptides works to stabilizing blood glucose.

Participants will:

* Take bitter melon peptides or a placebo every day for 12 weeks
* Visit the clinic on day 0, day 7, day 28 and day 84 for checkups and tests
* Glucose levels were monitored continuously by CGMs in the first 7 days and fasting blood samples were drawn at first visit (day0), third visit (day 28) and fourth visits (day 84)

ELIGIBILITY:
Inclusion Criteria:Participants were diagnosed with type 2 DM based on criteria recommended by the American Diabetes Association and required to have fasting plasma glucose of ≥126 mg/dl or an HbA1c of

≥ 6.5%, as measured on two separate occasions

Exclusion Criteria:cancer, active liver disease, current pregnancy , acute illness and autoimmune thyroid disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-27 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
glycemic variability | From enrollment (day0) to day7
  mean amplitude of glucose excursions and coefficient of variation, using CGM

SECONDARY OUTCOMES:
glycemic control | From enrollment (day0) to the end (day84)
  Glycated hemoglobulin A1C

OTHER OUTCOMES:
metabolic indicator | From enrollment (day0) to the end (day84)
  C-peptide